CLINICAL TRIAL: NCT03093571
Title: Auricular Acupuncture vs. Progressive Muscle Relaxation in Treatment of Pre-exam Anxiety - Randomised Crossover Study in Medical Students
Brief Title: Auricular Stimulation vs. Relaxation for Pre-exam Anxiety
Acronym: AAvsPMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BB 041/15
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auricular stimulation (Experimental): Auricular stimulation using indwelling auricular acupuncture needles
  Interventions: Device: Auricular stimulation
- Muscle relaxation (Experimental): Progressive muscle relaxation according to Jacobsen
  Interventions: Behavioral: Relaxation
- No intervention (No Intervention): No intervention, just monitoring of outcome parameters

INTERVENTIONS:
Device: Auricular stimulation — Auricular stimulation with indwelling fixed needles
  Arms: Auricular stimulation
Behavioral: Relaxation — Progressive muscle relaxation
  Arms: Muscle relaxation

SUMMARY:
Title of the study: Auricular acupuncture (AA) vs. progressive muscle relaxation for pre-exam anxiety - a randomised crossover study

Study period: 04 / 2015 - 07 / 2015

Principal Investigator: PD Dr. T. Usichenko Department of Anaesthesiology and Intensive Care, University Medicine of Greifswald

Aim of the study: To investigate the anxiolytic effect of AA vs. progressive muscle relaxation and vs. no intervention in students, passing the oral exams in anatomy at the University of Greifswald

Design: Prospective randomised crossover trial

Interventions: 1. AA using indwelling fixed needles, retained 24 h in situ 2. Progressive muscle relaxation

Number of volunteers: N = 30

Healthy medical students at the University of Greifswald Participants of the oral anatomy exams in spring/summer 2015 Without previous anxiolytic, sedative and analgesic medication No pregnancy or lactating Informed consent

Outcome measures: Anxiety level Heart rate, blood pressure Salivary α-amylase

ELIGIBILITY:
Inclusion Criteria:

1. Medical students at the University of Greifswald
2. Going to take part in oral exams of human anatomy
3. Participants without previous anxiolytic medication
4. Ability to understand and perform PMR
5. Written informed consent

Exclusion Criteria:

1. Recidivist alcoholics
2. Local auricular skin infection
3. Pregnant or lactating women
4. Participants with prosthetic or damaged cardiac valves, intracardiac and intravascular shunts, hypertrophic cardiomyopathy and mitral valve prolaps (risk of bacterial endocarditis according to guidelines of AHA)
5. Participants who are unable to understand the consent form
6. History of psychiatric disease

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Intensity of anxiety | 2 days
  State-trait-anxiety-inventory

SECONDARY OUTCOMES:
Salivary alpha-amylase | 1 day
  Enzymatic activity of salivary alpha-amylase
heart rate | 1 day
  heart rate
blood pressure | 1 day
  blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Klausenitz, MD. PhD, Principal Investigator — University Medicine of Greifswald

IPD SHARING:
Plan to Share IPD: Undecided